CLINICAL TRIAL: NCT02592382
Title: Nasal Xylitol for Recurrent Otitis Media
Brief Title: Nasal Xylitol in the Prevention of Otitis Media
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Carmel Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0429-13-rmb/CTIL
Record Dates: First submitted 2015-10-29; First posted 2015-10-30 (Estimated); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Otitis Media
MeSH Terms: conditions — Otitis Media

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Xylitol spray (Experimental): Xylitol nasal spray ( Xlear ltd which contains 10% of Xylitiol) given 3 times a day (one puff for each nostril) for three months period.
  Interventions: Dietary Supplement: Xylitol spray

INTERVENTIONS:
Dietary Supplement: Xylitol spray — xylitol nasal spray will be administered to this arm three times daily for three months

SUMMARY:
Acute otitis media (AOM) is one of the most prevalent and costly illnesses in children throughout the world. AOM can lead to chronic otitis media with effusion (OME) resulting in conductive hearing loss that can cause speech, language, academic, and social developmental delays.

Complementary and alternative medicines are being widely used for prevention of AOM.

Xylitol is a five carbon polyol (sugar alcohol) produced from natural plants and is used for preventing dental caries and AOM in children. It is commercially available in chewing gums, syrups and toothpastes washes, and other products. Xylitol was shown in several studies to prevent the culture of bacteria in the nasopharynx and oral cavity. It was proven to eliminate the ability of bacteria to attach to the mucosa of the upper respiratory system. It was proven to reduce the ability of bacteria to attach to the mucosa of the upper respiratory system. Previous study had shown that oral usage of Xylitol (as chewing gum or syrup) can reduce the incidence of rAOM by 30% as compared to placebo. But this treatment did not gain popularity since the initial clinical trial 30 years. There are several potential reasons for that. First, Xylitol should be administrated 5 times daily in order to be effective. Study that checked usage of oral Xylitol 3 times daily in children with rAOM did not find additional advantage as compared to placebo. Secondly, by using Xylitol orally we rely on the gut absorption and systemic distribution. Xylitol absorbs poorly in the gut and can cause some GI symptoms (like nausea and diarrhea) especially when used in a syrup (the preferred way in small children).

In this study the investigators aim to test the yield of Xylitol nasal spray as a preventive treatment in children with rAOM. By using Xylitol as nasal spray we deliver the active compound directly to the action site (nasopharynx- the AOM reservoir) and avoid the GI side effects

ELIGIBILITY:
Inclusion Criteria:

1. Children at the age of 1-5 years that suffered from recurrent otitis media (3 episodes in the last 6 months prior to entrance to the study)

Exclusion Criteria:

1. Children with immune deficiency
2. Children with craniofacial malformations
3. Children with chronic otitis media
4. Children that received prophylactic antibiotic treatment prior to entering the study (3 months )

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
prevalence of otitis media episodes | 6 months
  The number of events of acute otitis media during the study period of 6 months. The comparison is in 3 months intervals. pre-treatment, during treatment and post-treatment

SECONDARY OUTCOMES:
Side effects of treatment | 3 months
  any side effects of the treatment will be recorded

OTHER OUTCOMES:
Antimicrobial treatment | 9 months
  Collect the type (systemic or topical) of antimicrobial treatment prior and during the study
Parental diary | 6 months
  The parents will conduct a diary that will include AOM episodes, who made the diagnosis, what were the symptoms and what kind of treatment was given.

CONTACTS AND LOCATIONS:
Overall Officials: Arie Gordin, MD, Principal Investigator — Rambam Health Care Center
Locations (2):
- Israel (2):
  - Rambam Health Care Campus, Haifa
  - Carmel Medical Center, Haifa